CLINICAL TRIAL: NCT05809453
Title: Intranasal Cocaine and Temperature Regulation During Exercise
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU-2023-0094
Record Dates: First submitted 2023-03-16; First posted 2023-04-12 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Hyperthermia; Cocaine Use; Exercise
Keywords: thermoregulation; sweating; skin blood flow
MeSH Terms: conditions — Hyperthermia; Motor Activity | interventions — Cocaine; Lidocaine

STUDY DESIGN:
Intervention Model Description: We will conduct a double-blind, placebo-controlled, crossover study. Following informed consent and screening, eligible participants will be randomized to complete the cocaine or the lidocaine (placebo) trial first, with the other "agent" administered during the subsequent visit. During these experimental visits, we will first obtain "pre-drug" temperature and cardiovascular data, which will be followed by administer of cocaine or lidocaine intranasally. Participants will then enter the chamber set to warm environmental conditions. After further instrumentation in the warm environment, participants will perform mild to moderate intensity physical activity for 60 minutes. Throughout the 60 minutes of physical activity we will record body temperature and cardiovascular responses. Upon concluding the physical activity, subjects will rest while body temperature and cardiovascular responses are obtained post-physical activity.
Who Masked: Investigator
Masking Description: Our research nurse will know whether the participant will receive cocaine or lidocaine. All others involved in the protocol, including the participant, will not know which agent they received for which trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hot-Humid (Experimental): Participants will complete the trial in environmental conditions 38 degrees Celsius with 40% humidity.
  Interventions: Drug: Cocaine; Drug: Lidocaine
- Hot-Dry (Experimental): Participants will complete the trial in environmental conditions 41 degrees Celsius with 15% humidity.
  Interventions: Drug: Cocaine; Drug: Lidocaine

INTERVENTIONS:
Drug: Cocaine — Cocaine (cocaine hydrochloride 4% nasal solution) will be administered (3 mg/kg) intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise.
Drug: Lidocaine — Lidocaine (lidocaine hydrochloride 4% nasal solution) will be administered (3 mg/kg) intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise.

SUMMARY:
Assess the effects of intranasal cocaine on temperature regulation and whole-body sweat rate during exercise in warm environmental conditions.

DETAILED DESCRIPTION:
Previously it was shown that intranasal cocaine attenuates skin blood flow and sweating responses during passive heat stress, when compared to placebo. However, nothing is known about the effects of cocaine on whole-body temperature regulation during mild to moderate exercise in warm environmental condition.

This project will test the hypothesis that intranasal cocaine attenuates whole-body sweat rate, resulting in greater elevations in core temperature during mild to moderate exercise in warm environmental conditions.

Primary data include core temperature, skin temperatures, and whole body sweat rate. Secondary variables include cardiovascular responses, perceptions of exercise exertion and thermal comfort, and metabolic heat production. Intranasal lidocaine will be used as the placebo for cocaine. The selection of the drug administered during the first experimental trial will be randomized, with the other drug administered during the second experimental trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age
* Healthy
* Body mass index less than 31 kg/m^2
* Speak English
* Systolic blood pressure <140 mmHg
* Diastolic blood pressure <90 mmHg

Exclusion Criteria:

* Subjects not in the defined age range
* Participants who have cardiac, respiratory, neurological, and/or metabolic illnesses
* Any known history of renal or hepatic insufficiency/disease
* Pregnancy or breast feeding
* Body mass less than 60 kilograms
* Current smokers, as well as individuals who regularly smoked within the past 3 years
* Individuals with a history of drug abuse within the past 5 years
* Individuals who have an unexplained positive urine drug screen (e.g., some agents cause false-positive results and when agent abstained the drug screen is negative, one example could be an over the counter supplement)
* Currently taking pain modifying medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 participants who signed the consent were withdrawn from the study prior to visit 1 due to either elevated bp at screening visit or they started a new medication that disqualified them from participating in this study.
Groups:
- Hot-Humid: Cocaine First Then Lidocaine: Participants will complete two trials in environmental conditions 38 degrees Celsius with 40% humidity.
  Cocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 1. Lidocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 2.
- Hot-Humid: Lidocaine First Then Cocaine: Participants will complete two trials in environmental conditions 38 degrees Celsius with 40% humidity.
  Lidocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 1. Cocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 2.
- Hot-Dry: Cocaine First Then Lidocaine: Participants will complete 2 trials in environmental conditions 41 degrees Celsius with 15% humidity.
  Cocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 1. Lidocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 2.
- Hot-Dry: Lidocaine First Then Cocaine: Participants will complete 2 trials in environmental conditions 41 degrees Celsius with 15% humidity.
  Lidocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 1. Cocaine will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 2.
Period: Overall Study
Arm/Group | Hot-Humid: Cocaine First Then Lidocaine | Hot-Humid: Lidocaine First Then Cocaine | Hot-Dry: Cocaine First Then Lidocaine | Hot-Dry: Lidocaine First Then Cocaine
Started | 7 | 7 | 6 | 4
Completed | 6 | 7 | 6 | 4
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hot-Humid: Cocaine First Then Lidocaine | Hot-Humid: Lidocaine First Then Cocaine | Hot-Dry: Cocaine First Then Lidocaine | Hot-Dry: Lidocaine First Then Cocaine | Total
Number analyzed (Participants) | 6 | 7 | 6 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5) | 32 (3) | 28 (7) | 28 (4) | 30 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 1 | 11
  Male | 3 | 4 | 2 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 5 | 6 | 5 | 4 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 5 | 6 | 3 | 3 | 17
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Core Temperature
Description: Core temperature will be measured either from a temperature sensor pill or from a rectal temperature probe.
Time Frame: Core temperature is measured at baseline and at 60 minutes of heat exposure.
Measure: Mean (Standard Deviation); unit: Celsius
Groups:
- Hot-Humid: Cocaine; Hot-Humid: Lidocaine: Participants will complete two trials in environmental conditions 38 degrees Celsius with 40% humidity.
  Cocaine or lidocaine (randomized) will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 1. Cocaine or lidocaine (randomized) will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 2.
- Hot-Dry: Cocaine; Hot-Dry: Lidocaine: Participants will complete 2 trials in environmental conditions 41 degrees Celsius with 15% humidity.
  Cocaine or lidocaine (randomized) will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 1. Cocaine or lidocaine (randomized) will be administered intranasally prior to entering the warm environmental conditions and performing 60 minutes of exercise on visit 2.
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
Number analyzed (Participants) | 13 | 13 | 10 | 10
Celsius | 1.19 (0.32) | 1.09 (0.33) | 1.20 (0.27) | 0.89 (0.23)

2. Secondary Outcome: End Skin Temperature
Description: Skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin
Time Frame: Measured at the end of heat exposure, 90 minutes from cocaine/lidocaine administration
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
Number analyzed (Participants) | 13 | 13 | 10 | 10
Celsius | 35.83 (0.44) | 35.57 (0.59) | 35.80 (0.81) | 35.39 (0.99)

3. Secondary Outcome: End Heart Rate
Description: Heart rate will be measured from ECG electrodes attached to the participant
Time Frame: Measured at the end of heat exposure, 90 minutes from Cocaine/ lidocaine administration
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
Number analyzed (Participants) | 13 | 13 | 10 | 10
BPM | 151 (21) | 147 (18) | 147 (20) | 134 (18)

4. Secondary Outcome: Whole Body Sweat Rate
Description: Whole body sweat rate is calculated by subtracting the participants post-heat exposure nude body weight from their pre-heat exposure nude body weight
Time Frame: Within 30 minutes before exposure to warm environmental conditions (before cocaine/ lidocaine administration) and immediately after the heat exposure (90 minutes post cocaine/ lidocaine administration)
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
Number analyzed (Participants) | 13 | 13 | 10 | 10
L/hour | 0.83 (0.25) | 0.79 (0.27) | 0.79 (0.15) | 0.84 (0.15)

5. Secondary Outcome: End Mean Arterial Pressure
Description: Systolic and diastolic blood pressure will be measured from a cuff placed on the upper arm.
Time Frame: Measured at the end of heat exposure, 90 minutes from cocaine/ lidocaine administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
Number analyzed (Participants) | 13 | 13 | 10 | 10
mmHg | 85 (7) | 89 (8) | 86 (10) | 87 (9)

6. Secondary Outcome: End Thermal Sensation
Description: Subjective assessment of how hot the subject feels.
  Title of Scale: Thermal Sensation Scale; Minimum value: -50 "unbearably cold"; Maximum value: 50: "unbearably hot" Scale presents numbers in increments of 5
Time Frame: These values will be obtained at end of the 60 minute heat exposure (90 minutes post cocaine/ lidocaine administration)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
Number analyzed (Participants) | 13 | 13 | 10 | 10
units on a scale | 31 (14) | 37 (9) | 26 (12) | 27 (15)

ADVERSE EVENTS:
Time Frame: Adverse data was collected through study completion, an average of one month.
Arm/Group | Hot-Humid: Cocaine | Hot-Humid: Lidocaine | Hot-Dry: Cocaine | Hot-Dry: Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT05809453/Prot_SAP_000.pdf